CLINICAL TRIAL: NCT04674436
Title: Can a 6-minute Walking or Resting Break Improve Executive Function and Gaming
Brief Title: Can a 6-minute Walking or Resting Break Improve Executive Function in Gamers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Joanne DiFrancisco-Donoghue, Associate Professor, New York Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1566
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6 minute walking break (Experimental): Participants will walk casually for 6 minutes following one hour of game play, then continue play for one more hour.
  Interventions: Behavioral: Walking
- 6 minute rest break (Experimental): Participants will rest supine for 6 minutes following one hour of game play, then continue play for one more hour.
  Interventions: Behavioral: Walking
- Continuous play (No Intervention): Participants will play continuous for 2 hours.

INTERVENTIONS:
Behavioral: Walking — 6 minute casual walk
  Arms: 6 minute rest break; 6 minute walking break

SUMMARY:
This study will ask ranked first person shooters in esports to participate on three separate days from their home computer to test executive function prior tp play and following two hours of play. One testing day will incorporate a 6 minute walk break, another day will incorporate a 6 minute rest break, and the third day will be continuous play. Executive tests will be administered electronically prior to game play and post game play.

DETAILED DESCRIPTION:
A ranked first person shooter player will play for two hours each session, and on separate days will take a 6 minute walking break or a 6 minute resting break within 2 hours of game play. This study is virtual and you may play from your regular home gaming computer. The third day will be continuous play.

The study will take place on 3 separate days. Preferably 2 -3 days in -between testing days.

* Participants will sign an electronic consent form to sign and agree to participate. It will explain the study in detail.
* Participants will then be asked to take two executive function tests online. These test will be sent electronically through email. This is for practice. These tests take approximately 6-7 minutes.
* We will schedule one day where the participant will play a first -person shooter game. Prior to playing the participants will be take to take the two executive function tests.
* On one day the participant will be asked to stop after the first hour (they will be allowed to finish the test) they will either walk for 6 minutes near their computer or rest for 6 minutes. Participants will be contacted through cell phones or discord.
* Game play will resume normally for another hour. When that hour is completed the participant will be asked to take the two online tests again.
* This will be 2 days. The third day the participant will take the online tests and play continuous for 2 hours with no break and then repeat the online tests.

ELIGIBILITY:
Inclusion Criteria:1. Women or men 18-25 years of age 2. Play first-person shooter games with a ranking of "gold" or higher (self reported).

-

Exclusion Criteria:1. Any participants that do not have a competitive ranking 2. Any participants that are colorblind (self reported) 3. Any participants that have sustained previous hand injuries within the last year, or suffer from chronic wrist pain.

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Executive Function | 2 hours
  The primary purpose of this study is to evaluate executive function changes following a 6-minute walking break to a 6 minute resting break in competitive esport players following 60 minutes of prolonged play

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donoghue, Principal Investigator — New York Institute of Technology
Locations (2):
- United States (2):
  - New York Institute of Technology College of Osteopathic Medicine, Old Westbury, New York
  - New York Institute of Technology, Old Westbury, New York

IPD SHARING:
Plan to Share IPD: No